CLINICAL TRIAL: NCT00597688
Title: Oral Mucosal Decontamination With Chlorhexidine for Prevention of Ventilator Associated Pneumonia in Children - A Randomized Controlled Trial
Brief Title: Role of Oral Chlorhexidine Gel in Prevention of Ventilator Associated Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Meghna Raju Sebastian, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Meghna
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2009-02

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Chlorhexidine gel
  Interventions: Drug: Chlorhexidine gel
- 2 (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: Chlorhexidine gel — Oral mucosal application of chlorhexidine gel
  Arms: 1
Drug: Placebo gel — Oral mucosal application of placebo gel
  Arms: 2

SUMMARY:
The purpose of this study is to determine if oral mucosal application of chlorhexidine gel will prevent the development of ventilator associated pneumonia in children.

DETAILED DESCRIPTION:
Ventilator associated pneumonia as the name suggests refers to pneumonia occurring in the setting of mechanical ventilation. It accounts of 86% of nosocomial pneumonia and in contrast to other more common nosocomial infections is accompanied by a mortality rate of upto 76% in certain settings. A number of preventive methods have been studied to reduce the rate of VAP but a consensus is lacking with regards to appropriate preventive strategies. Studies in adults have shown a beneficial effect of oral mucosal application of chlorhexidine but similar studies in pediatric population are not available. This research project aims at addressing the gap.

ELIGIBILITY:
Inclusion criteria:

1. Patients in PICU requiring mechanical ventilation
2. Above the age of 3 months
3. Oro or nasotracheal intubation

Exclusion criteria:

1. Known hypersensitivity to chlorhexidine
2. Inability to access the oral cavity for any reason
3. Patients with tracheostomy
4. Mechanical ventilation for more than 24 hours prior to PICU admission.
5. Death or extubation within 24 hours of ICU admission.

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of ventilator associated pneumonia as defined by CDC diagnostic criteria | 21 days

SECONDARY OUTCOMES:
Antibiotic sensitivity of organism cultured | 21 days
Duration of hospital stay | 21 days
Duration of ICU stay | 21 days
In hospital mortality rate | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: RAKESH LODHA, Study Director — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Sebastian MR, Lodha R, Kapil A, Kabra SK. Oral mucosal decontamination with chlorhexidine for the prevention of ventilator-associated pneumonia in children - a randomized, controlled trial. Pediatr Crit Care Med. 2012 Sep;13(5):e305-10. doi: 10.1097/PCC.0b013e31824ea119. PMID 22760426